CLINICAL TRIAL: NCT05369949
Title: Effect of DEXmedetomidine and LOw Dose Sevoflurane on the Release of Serum Neurofilament Light in Congenital Cardiac Surgery.
Brief Title: DEX vs SEVO in Congenital Heart Surgery
Acronym: DEXLOSNeuro
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mona Momeni, MD, PhD, Deputy Anesthesiologist in Chief. MD,PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ethical Advice
Record Dates: First submitted 2022-04-21; First posted 2022-05-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-07

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The Intervention Drug is DEXMEDETOMIDINE
Masking Description: The patient's parents will be informed of the study allocation in case they wish to know this, otherwise they are not supposed to be aware of group allocation. Persons who will assess the neurodevelopment outcome will not be aware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Experimental): Participants will receive an intraoperative and postoperative DEX infusion. In addition a low dose of sevoflurane will be administered.
  Interventions: Drug: DEX group
- Control group (Active Comparator): Participants will receive general anesthesia with sevoflurane according to institutinal's practice.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: DEX group — Participants will receive a dexmedetomidine infusion in addition to low dose sevoflurane anesthesia.
  Arms: DEX group
Other: Control group — Participants will receive general anesthesia based on institutional's practice with commonly used doses of sevoflurane.
  Arms: Control group

SUMMARY:
Anesthesia-related neurotoxicity in the developing brain is still a concern although evidence in humans is debatable. Moreover, it is unclear whether repeated and/or prolonged exposures are harmless and whether their effects are more pronounced in newborns and infants with brains more vulnerable to injury. One such specific group of patients is children with congenital heart disease (CHD). Nearly, half of the school-age survivors with CHD exhibit neurodevelopmental symptoms. It is thus important to elucidate whether any plausible neurotoxicity of the commonly used anesthetic agents can be observed in this population, and whether specific neuroprotective strategies can be demonstrated within the frame of a randomized controlled trial (RCT).

Animal data have shown that dexmedetomidine (DEX) induces neuroprotective effects only at well-adjusted doses. One major issue with trials of anesthetic neurotoxicity is the latency between the conduct of these studies and the assessment of neurodevelopmental outcome. In contrast, the use of biomarkers of neuronal injury could be extremely valuable. Serum Neurofilament Light (NfL) has been shown to be a sensitive and specific marker of neuronal injury and is associated with neurologic outcome of children with various pathologies. The investigators hypothesize that in congenital heart surgery, use of DEX as main anesthetic agent in conjunction with low dose sevoflurane results in less release of serum NfL and is thus potentially less neurotoxic compared to the current standard of care. The hypothesis is tested with a RCT including patients between 0 - 3y undergoing surgery with cardiopulmonary bypass. To avoid any neurotoxicity due to anesthetic overdose, intraoperative burst suppression will be avoided. In addition to postoperative comparison of serum NfL, postoperative electroencephalogram and neurodevelopmental outcome of both groups will be compared taking into consideration the genetic background.

ELIGIBILITY:
Inclusion Criteria:

* Patients up to 3 years
* Must undergo cardiac surgery with CPB

Exclusion Criteria:

* Preoperative chronic kidney disease (glomerular filtration rate of less than 30 ml/min per 1.73m2 for greater than 3 months)
* Preoperative cerebral hemorrhage, stroke or
* Preoperative seizures
* Abnormal preoperative cerebral ultrasound
* Preoperative Extracorporeal Life Support
* Preoperative sedated and intubated patients
* Preterm newborns (< 32 W gestational age)
* Newborns weighing < 2 kg
* Patients with Williams-Beuren syndrome.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-01-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum Neurofilament Light | At 24 hours postoperatively
  To show a difference of change in serum NfL concentrations between both groups at 24h compared to baseline values.

SECONDARY OUTCOMES:
Concentration of serum Neurofilament Light | Baseline before start of anesthesia
Concentration of serum Neurofilament Light | Start of cardiopulmonary bypass
Concentration of serum Neurofilament Light | At 72 hours postoperatively
Concentration of serum Neurofilament Light | At postoperative day 5
Neurodevelopmental outcome testing | 3 months postoperatively
  Bailey Scales of Infant and Toddler Development - Third Edition. Higher scores are better.
Neurodevelopmental outcome testing | 6 months postoperatively
  Bailey Scales of Infant and Toddler Development - Third Edition. Higher scores are better.
Postoperative electroencephalogram registration | 24 hours
  Number of seizures
Dose of Analgesics | 72 hours postoperatively
  Use and dose of analgesics
Renal function | 7 days postoperatively
  Defined by pediatric RIFLE criteria
Concentration of regional cerebral oxygenation | Intraoperatively
  Area Under Curve of time spent below rSO2 levels of 50%; Area Under Curve of time spent below baseline rSO2 levels
Postoperative electroencephalogram registration | 24 hours
  Number of burst-suppression episodes
Postoperative electroencephalogram registration | 24 hours
  Duration of burst-suppression episodes
Postoperative electroencephalogram registration | 24 hours
  Duration of seizures
Time of exsudation | 7 days postoperatively
  time to extubation
Pediatric Intensive Care Unit stay | Up to 24 weeks
  Duration of stay in Pediatric Intensive Care Unit
Hospital stay | Up to 24 weeks
  Days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mona Momeni, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No